CLINICAL TRIAL: NCT00748865
Title: Acute Comfort and Blur of Systane Ultra and Systane
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: M-08-09
Record Dates: First submitted 2008-09-05; First posted 2008-09-09 (Estimated); Results first posted 2010-03-11 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Dry Eye
Keywords: Dry Eye; Artificial Tears
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Systane Ultra (Experimental): Systane Ultra 1 drop each eye one time
  Interventions: Other: Systane Ultra Lubricant Eye Drops
- Systane (Active Comparator): Systane 1 drop each eye one time
  Interventions: Other: Systane Lubricant Eye Drops

INTERVENTIONS:
Other: Systane Ultra Lubricant Eye Drops — Systane Ultra Lubricant Eye Drops 1 drop each eye one time
  Arms: Systane Ultra
Other: Systane Lubricant Eye Drops — Systane Lubricant Eye Drops 1 drop each eye one time
  Arms: Systane

SUMMARY:
To evaluate drop comfort, acceptability, preference and blue profile between two marketed artificial tears in both dry eyes and non-dry eye patient population.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of dry eye

Exclusion Criteria:

* Use of contact lens within 7 days preceding enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-07; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center for Trial Location, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20 dry eye subjects
Pre-assignment Details: Randomized, double-masked, cross-over design
Groups:
- Systane Ultra Drops, Then Systane Drops: Patients received Systane Ultra Drops first, then received Systane Drops.
- Systane Drops, Then Systane Ultra Drops: Patients first received Systane Drops, then received Systane Ultra Drops
Period: Overall Study
Arm/Group | Systane Ultra Drops, Then Systane Drops | Systane Drops, Then Systane Ultra Drops
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Drop Comfort
Description: Drop comfort grading scale is a 0 to 9 scale, with 0 meaning most comfortable and 9 meaning most uncomfortable,
Time Frame: once upon instillation
Measure: Median (Standard Deviation); unit: Units on a scale
Groups:
- Systane Ultra: Systane Ultra
- Systane: Systane
Arm/Group | Systane Ultra | Systane
Number analyzed (Participants) | 20 | 20
Units on a scale | 0.55 (0.69) | 0.60 (0.68)

ADVERSE EVENTS:
Arm/Group | Systane Ultra | Systane
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI should hold confidential, and not disclose directly or indirectly to any third party other than Contractors, the data arising out of the study. Alcon reserves the right of prior review of any publication or presentation of information related to the study.